CLINICAL TRIAL: NCT01983228
Title: A Proactive Walking Trial to Reduce Pain in Black Veterans
Acronym: ACTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 13-030
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Musculoskeletal Pain
Keywords: Musculoskeletal Pain; Walking; African American; Telephone Coaching; Pedometer
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Intervention participants will receive a pedometer-mediated walking intervention that will incorporate Action Planning and the use of MI and CBT techniques. The intervention will be delivered in 6 telephone counseling sessions over three months.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Usual Care (No Intervention): Participants randomized to the usual care control condition will receive pedometers and an informational brochure.
- Arm 2: Intervention Group (Experimental): Participants assigned to the intervention group will receive personalized recruitment materials, including a letter and brochure describing the program and the benefits of walking for pain. They will also receive pedometers. Participants will complete 6 sessions of telephone coaching over a 10-12 week period, using a patient workbook with visual aids (e.g., diagram of the pain/inactivity cycle) and worksheets that they will complete during the counseling sessions. Participants are expected to receive approximately 180 minutes of total therapist time during the study.
  Interventions: Behavioral: Intervention Condition

INTERVENTIONS:
Behavioral: Intervention Condition — Intervention participants will complete 6 sessions of telephone coaching over a 10-12 week period, using a patient workbook with visual aids (e.g., diagram of the pain/inactivity cycle) and worksheets that they will complete during the counseling sessions. Participants are expected to receive approximately 180 minutes of total therapist time during the study.
  Arms: Arm 2: Intervention Group

SUMMARY:
The long term goal is to improve the quality and equity of chronic pain treatment among VA patients. The primary objective of this study is to improve pain outcomes among black VA patients with chronic, musculoskeletal (MSK) pain, who experience poorer pain treatment and outcomes than their white counterparts. The work proposed is expected to result in a non-pharmacological intervention, delivered by telephone, designed to reduce pain and improve functioning among black patients with MSK pain, by promoting walking. This intervention is specifically designed to address factors that contribute to MSK pain among black Veterans; however, the investigators expect that it will also benefit non-black Veterans. The proposed research is innovative, in its use of proactive outreach and recent advances in self-regulation strategies (such as Action Planning) to help black Veterans overcome psychological, environmental, utilization-related, and provider-related barriers that contribute to pain.

DETAILED DESCRIPTION:
BACKGROUND/RATIONALE:

Chronic musculoskeletal (MSK) pain is one of the most common conditions among Veterans, affecting approximately 60% of those seen in VA primary care. Although perceived effectiveness of chronic pain treatment is low among all VA patients, black patients are less likely than whites to perceive their treatment as effective, and are more likely to experience functional limitations due to pain. There is growing consensus that chronic pain is best addressed by a biopsychosocial approach that acknowledges the role of psychological and environmental contributors to pain, some of which differ by race and hence contribute to disparities. For example, blacks experience greater pain-related fear and lower self-efficacy in coping with pain (psychological contributors), and neighborhoods that make physical activity difficult (environmental contributors). However, there is a lack of effective interventions to improve pain treatment among minority patients, particularly those that target psychological and environmental contributors.

OBJECTIVES:

The long term goal is to improve the quality and equity of pain treatment in order to improve pain outcomes for all Veterans. The objective of this application is to test the effectiveness of a multi-component intervention that specifically targets known barriers to effective pain care among black Veterans with chronic MSK pain. The primary hypothesis is that a telephone-delivered intervention, which emphasizes walking and incorporates Action Planning, Motivational Interviewing (MI) and Cognitive Behavioral Therapy (CBT) techniques, and the use of pedometers, will improve core chronic pain outcomes in black Veterans. Secondarily, we will determine whether our intervention also benefits non-black patients with MSK.

METHODS:

The investigators propose a randomized trial to test the effectiveness of the intervention compared with usual care (UC) among 500 patients with chronic MSK pain, with a minimum of 250 Black participants. Patients from the Atlanta VAMC will be identified using administrative data. Patients will be screened by phone, and, if eligible, will be mailed the baseline survey to complete and mail back. Eligible patients who complete the baseline survey will be randomly assigned to the usual care (UC) or intervention condition (IC). Intervention participants will receive a pedometer-mediated walking intervention that will incorporate Action Planning and the use of MI and CBT techniques. The intervention will be delivered in 6 telephone counseling sessions over three months. Patients in the UC condition will receive an informational brochure and a pedometer. The study is powered to find a difference between the IC and UC groups within the black and non-black groups. The primary outcome is chronic pain-related physical functioning, assessed by the revised Roland and Morris Disability Questionnaire, a measure recommended by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT). We will also examine whether the intervention improves other IMMPACT-recommended domains (pain intensity, emotional functioning, and ratings of overall improvement). Secondary objectives include examining potential mediators targeted by the intervention, exploring whether the intervention affects service utilization and use of opioid analgesics, and exploring whether the intervention reduces racial disparities in pain outcomes. Measures will be assessed by mail and phone survey at baseline, 3 months, and 6 months. Data analysis of primary aims will follow intent-to-treat methodology.

FINDINGS:

None at this time.

STATUS:

Focus groups were conducted at the Atlanta VAMC in September and October 2015. These focus groups provided valuable information that led us to refine our recruitment materials. Focus groups also yielded important information for our counselors, including potential communication barriers and barriers to walking. During January - April 2016, we conducted a pilot test of our intervention with 3 participants. We began the trial on July 2016. Recruitment and randomization were completed in June 2019. The intervention activities were completed in September 2019. Follow-up survey data collection is currently ongoing.

IMPACT:

The work proposed is expected to result in a non-pharmacological intervention, delivered by telephone, designed to reduce pain and improve functioning among black patients with MSK pain, by promoting walking.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must receive care at the Atlanta VAMC and
* have back, hip or knee pain for a duration of at least 6 months,
* moderate-severe pain intensity and interference with function (defined as a PEG score of 5 or greater),
* self-reported ability to walk at least 1 block, and
* must be able to communicate effectively by telephone (no cognitive disability). The investigators will not exclude patients who are on medication or receiving interventions to treat their chronic pain. The investigators will include the approximately 10% of patients who have no race data; race data will be collected on the brief screening survey.

Exclusion Criteria:

The investigators will not include any vulnerable populations or those who meet any of the following exclusion criteria that may interfere with the outcome assessment: a) moderately severe cognitive impairment defined as > 2 errors on a brief cognitive screener; b) anticipated back, knee, hip, or other major surgery within the next 6 months; c) patients who say they are unable to walk at least a block; d) patients who say they would be unavailable to participate in a 6 month study; e) patients with active psychotic symptoms, suicidality, and/or active manic episode or poorly controlled bipolar disorder, as determined by chart review.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana J. Burgess, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhimani RH, Cross LJ, Taylor BC, Meis LA, Fu SS, Allen KD, Krein SL, Do T, Kerns RD, Burgess DJ. Taking ACTION to reduce pain: ACTION study rationale, design and protocol of a randomized trial of a proactive telephone-based coaching intervention for chronic musculoskeletal pain among African Americans. BMC Musculoskelet Disord. 2017 Jan 13;18(1):15. doi: 10.1186/s12891-016-1363-6. PMID 28086853
- [Result] Burgess DJ, Hagel Campbell E, Hammett P, Allen KD, Fu SS, Heapy A, Kerns RD, Krein SL, Meis LA, Bangerter A, Cross LJS, Do T, Saenger M, Taylor BC. Taking ACTION to Reduce Pain: a Randomized Clinical Trial of a Walking-Focused, Proactive Coaching Intervention for Black Patients with Chronic Musculoskeletal Pain. J Gen Intern Med. 2022 Nov;37(14):3585-3593. doi: 10.1007/s11606-021-07376-2. Epub 2022 Feb 7. PMID 35132545
- [Result] Hammett PJ, Eliacin J, Makris UE, Allen KD, Kerns RD, Heapy A, Goldsmith ES, Meis LA, Taylor BC, Saenger M, Cross LJS, Do T, Branson M, Burgess DJ. An Analysis of the Role of Mental Health in a Randomized Trial of a Walking Intervention for Black Veterans With Chronic Pain. J Pain. 2023 Jan;24(1):55-67. doi: 10.1016/j.jpain.2022.07.002. Epub 2022 Sep 23. PMID 36162790
- [Derived] Hammett PJ, Eliacin J, Saenger M, Allen KD, Meis LA, Krein SL, Taylor BC, Branson M, Fu SS, Burgess DJ. The Association Between Racialized Discrimination in Health Care and Pain Among Black Patients With Mental Health Diagnoses. J Pain. 2024 Jan;25(1):217-227. doi: 10.1016/j.jpain.2023.08.004. Epub 2023 Aug 15. PMID 37591480

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Started | 249 | 251
Completed | 211 | 189
Not Completed | 38 | 62

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Usual Care: Participants randomized to the usual care control condition received a pedometer and an informational brochure about the benefits of walking. They were instructed to use and record their steps with the pedometer the week before the baseline survey and the follow-up surveys.
- Arm 2: Intervention Group: Intervention participants received a pedometer and tailored materials (a letter and brochure) describing the program and the benefits of walking and physical activity to help manage pain. The manualized, ACTION intervention consisted of six 30- to 60-minute long telephone coaching sessions over an 8-14-week period, delivered by counselors trained in motivational interviewing. Participants were coached to create and write action plans for their proposed walking activity, during the week(s) between coaching sessions, using templates contained in their workbooks. Counselors were also trained to help participants develop specific types of action plans to overcome barriers, strengthen helpful factors, and involve friends and family members. Pedometers were used as a tool to promote walking through feedback, goal setting, and monitoring.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group | Total
Number analyzed (Participants) | 249 | 251 | 500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 166 | 170 | 336
  >=65 years | 83 | 81 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (10.9) | 59.6 (11.1) | 59.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 58 | 124
  Male | 183 | 193 | 376
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 241 | 248 | 489
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 249 | 251 | 500

OUTCOME MEASURES:

1. Primary Outcome: 30% Improvement in Physical Functioning as Assessed by the Roland Morris Disability Questionnaire [RMDQ]) at 6 Months
Description: 30% improvement on the Roland Morris Disability Questionnaire [RMDQ]) from baseline over the 6-month follow-up period.
  Minimum value: 0. Maximum value: 11. Higher scores indicate greater disability.
Time Frame: Assessed at baseline and 6 months
Population: Primary Analysis completed in Black participants only.
Measure: Number; unit: participants w/ >= 30% improvement
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 154 | 142
participants w/ >= 30% improvement | 38 | 46
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; measured change as a responder yes/no (30% or greater improvement from baseline); Test type: Superiority; p = 0.09, Regression, Logistic — Multiple logistic regression adjusted for use of walking aids and opioids (both significantly difference between arms at baseline); Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.94 to 2.77]

2. Secondary Outcome: Change in Brief Pain Intensity Scale at 6 Months
Description: Pain intensity assessed by change in Brief Pain Intensity Scale at 6 months. Min=0, max=10, higher scores indicate worse outcome. The investigators will assess change in this outcome from baseline to 6 months.
Time Frame: Baseline and 6 months
Population: Analysis completed in Black participants only
Measure: Mean (Standard Error); unit: change in score on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
change in score on a scale | -0.24 (0.14) | -0.45 (0.15)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.34, Regression, Linear — Multiple linear regression adjusted for use of walking aids and opioids (both significantly difference between arms at baseline); Median Difference (Final Values) = -0.20, 95% CI 2-sided [-0.62 to 0.21]

3. Secondary Outcome: Change in Generalized Anxiety Disorder at 6 Months
Description: Change in Generalized Anxiety Disorder assessed by 7-item Generalized Anxiety Disorder scale (GAD-7) Min=0, max=21, higher scores indicate worse outcome. The investigators will assess change in this outcome from baseline to 6 months.
Time Frame: Baseline and 6 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: change in score on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
change in score on a scale | -0.43 (0.41) | -0.95 (0.43)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.38, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.69 to 0.65]

4. Secondary Outcome: Change in Depression at 6 Months
Description: Change in Depression at 6 months assessed by 8-item Patient Health Questionnaire (PHQ-8).
  Min=0, max=24, higher scores indicate worse outcome. The investigators will assess change in this outcome from baseline to 6 months.
Time Frame: Baseline and 6 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: change in score on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
change in score on a scale | -0.96 (0.38) | -1.56 (0.40)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.28, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-1.68 to 0.49]

5. Secondary Outcome: Overall Improvement Assessed by Patient Global Impression of Change Scale at 6 Months
Description: Single item measure of patient global impression of change. The investigators will assess this outcome at 6 months. Min=1, max=7, higher scores indicate worse outcome.
Time Frame: 6 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
units on a scale | 3.87 (0.14) | 4.26 (0.13)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.05, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.00 to 0.77]

6. Secondary Outcome: Mean Change in Average Daily Total Steps at 6 Months
Description: Pedometer data recorded over past 7 days on patient logs The investigators will assess mean change in this outcome from baseline to 6 months.
Time Frame: baseline and 6 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: change in number of steps
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
change in number of steps | 397.21 (220.03) | 591.11 (243.02)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority — Multiple linear regression adjusted for use of walking aids and opioids (both significantly difference between arms at baseline); p = 0.56, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 193.90, 95% CI 2-sided [-454.93 to 842.73]

7. Secondary Outcome: 30% Improvement in Physical Functioning as Assessed by the Roland Morris Disability Questionnaire [RMDQ]) at 3 Months
Description: 30% improvement on the Roland Morris Disability Questionnaire [RMDQ]) from baseline over the 3-month follow-up period.
  Minimum = 0 Maximum = 11 Higher scores indicate greater disability The investigators will assess change in this outcome from baseline to 3 months.
Time Frame: Baseline and 3 months
Population: Analysis completed in Black participants only.
Measure: Number; unit: participants w/ >= 30% improvement
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 149 | 139
participants w/ >= 30% improvement | 34 | 40
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; measured change as a responder yes/no (30% or greater improvement from baseline); Test type: Superiority; p = 0.16, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.85 to 2.62]

8. Secondary Outcome: Change in Brief Pain Intensity Scale at 3 Months
Description: Pain intensity assessed by Brief Pain Intensity Scale Min=0, max=10, higher scores indicate worse outcome. The investigators will assess change in this outcome from baseline to 3 months.
Time Frame: Baseline and 3 months
Population: Analysis completed in Black participants only
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
units on a scale | 0.02 (0.14) | -0.58 (0.15)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.002, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.99 to -0.23]

9. Secondary Outcome: Change in Generalized Anxiety Disorder, at 3 Months
Description: Change in Generalized Anxiety Disorder (GAD-7). Min=0, max=21, higher scores indicate worse outcome. The investigators will assess change in this outcome from baseline to 3 months.
Time Frame: Baseline and 3 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
units on a scale | -0.75 (0.42) | -0.39 (0.44)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.54, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [-0.79 to 1.51]

10. Secondary Outcome: Change in Depression Using 3 Month
Description: Change in Depression at 3 months using the 8-item Patient Health Questionnaire (PHQ-8) Min=0, max=24, higher scores indicate worse outcome. The investigators will assess change in this outcome from baseline to 3 months.
Time Frame: Baseline and 3 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
units on a scale | -1.27 (0.42) | -0.79 (0.43)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.41, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-0.66 to 1.62]

11. Secondary Outcome: Overall Improvement Assessed by Patient Global Impression of Change Scale at 3 Months
Description: Single item measure of patient global impression of change. The investigators will assess this outcome using the 3-month assessment. Min=1, max=7, higher scores indicate worse outcome
Time Frame: 3 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
units on a scale | 4.51 (0.13) | 3.79 (0.13)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p < 0.0001, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-1.07 to -0.38]

12. Secondary Outcome: Mean Change in Average Daily Total Steps, at 3 Months
Description: Pedometer data recorded over past 7 days on patient logs. The investigators will assess mean change in this outcome from baseline to 3 months.
Time Frame: 3 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: change in number of steps
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
change in number of steps | 92.97 (207.63) | 633.75 (219.56)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.06, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 540.78, 95% CI 2-sided [-28.77 to 1110.33]

13. Other Pre Specified Outcome: Pain Self-efficacy Questionnaire (PSEQ) at 6 Months
Description: Pain self-efficacy questionnaire (PSEQ) at 6 months Min: 10; Max: 60 Higher scores reflect stronger self-efficacy beliefs
Time Frame: 6 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
score on a scale | 32.22 (1.08) | 35.15 (1.09)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.05, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 2.93, 95% CI 2-sided [-0.01 to 5.86]

14. Other Pre Specified Outcome: Exercise Self-efficacy- Exercise Regularity Scale at 6 Months
Description: Exercise self-efficacy and regularity scale at 6 months Min=1, max=10, higher scores indicate better outcome.
Time Frame: 6 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
score on a scale | 4.45 (0.22) | 5.21 (0.23)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.01, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [0.15 to 1.36]

15. Other Pre Specified Outcome: Pain-related Fear Avoidance: Fear-Avoidance Beliefs Questionnaire (FABQ) Scale 1 at 6 Months.
Description: Pain-related Fear Avoidance: Fear-Avoidance Beliefs Questionnaire (FABQ) Scale 1 at 6 months.
  Min=0, max=24, higher scores indicate worse outcome.
Time Frame: 6 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
score on a scale | 16.23 (0.53) | 15.17 (0.55)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.15, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-2.53 to 0.39]

16. Other Pre Specified Outcome: Marcus Social Support Questions
Description: Family Social Support for Exercise at 6 months Min: 0 Max: 40 Higher scores indicate greater social support.
Time Frame: 6 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
score on a scale | 10.37 (0.41) | 10.70 (0.43)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.56, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.80 to 1.47]

17. Other Pre Specified Outcome: Service Utilization Treatment Quality at 6 Months
Description: Rating of quality of pain care received at the VA. Scale 1 (poor) to 5 (excellent)
Time Frame: 6 months
Population: Analysis completed in Black participants only.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
units on a scale | 2.75 (0.11) | 2.89 (0.12)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.38, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.17 to 0.46]

18. Other Pre Specified Outcome: Opioid Use for Pain Treatment at 6 Months
Description: Use of Opioids for pain treatment - Yes/No.
Time Frame: 6 months
Population: Analysis completed in Black participants only.
Measure: Number; unit: participants who reported using Opioids
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 154 | 143
participants who reported using Opioids | 79 | 80
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.56, Regression, Logistic — Logistic regression modeling the odds of yes to using opioids for pain treatment adjusting for use of walking aids and opioids (both significantly difference between arms at baseline); Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.66 to 2.19]

19. Other Pre Specified Outcome: Subjective Social Status
Description: Ladder representing subjective social status Min: 1; Max: 10 Higher numbers indicated greater subjective social status
Time Frame: 3 months
Population: Analysis completed in Black participants only
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
Number analyzed (Participants) | 193 | 187
units on a scale | 5.13 (0.19) | 5.47 (0.19)
Statistical Analysis 1: Comparison: Arm 1: Usual Care vs Arm 2: Intervention Group; Test type: Superiority; p = 0.21, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.18 to 0.84]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from September 2016 when intervention began through February 2020 when follow-up data collection ended. This is equal to 3 years and 5 months.
Arm/Group | Arm 1: Usual Care | Arm 2: Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/250
Serious Adverse Events (participants affected / at risk) | 0/249 | 0/250
Other Adverse Events (participants affected / at risk) | 0/249 | 0/251

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT01983228/Prot_SAP_000.pdf